CLINICAL TRIAL: NCT07397143
Title: Biomechanical Simulation Analysis of the Lower Extremity During Running in Males With Type A Lower Crossed Syndrome.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Shazlin Shaharudin, Associate Professor, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USM/JEPeM/KK/24090808
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-12

CONDITIONS: Lower Crossed Syndrome
Keywords: Lower Crossed Syndrome; Exercise Intervention; Kettlebell Training; Postural Imbalance; Muscle Imbalance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention Group (Experimental): Participants in this group perform a structured, supervised kettlebell-based exercise program three times per week for a duration of eight weeks.
  Interventions: Other: Kettlebell Exercise Program
- Control Group (No Intervention): Participants in this group receive usual care and do not participate in the exercise intervention during the study period.

INTERVENTIONS:
Other: Kettlebell Exercise Program — A structured, supervised kettlebell-based exercise program performed three times per week for eight weeks. Each session lasts approximately 40 minutes and includes warm-up, kettlebell exercises targeting core and lower limb muscles, and cool-down. The program is designed to improve muscle balance and postural control in male patients with Type A Lower Crossed Syndrome .
  Other Names: Structured Kettlebell Training
  Arms: Exercise Intervention Group

SUMMARY:
This study aims to examine the effects of an 8-week exercise program on male patients with lower crossed syndrome type A. Participants are randomly assigned to either an exercise group or a control group. The exercise group takes part in a supervised kettlebell-based exercise program three times per week for eight weeks, while the control group receives usual care without the exercise program. Measurements are taken before and after the intervention to compare changes between the two groups.

DETAILED DESCRIPTION:
This randomized controlled study investigates the effects of an exercise intervention on male patients with lower crossed syndrome type A. Participants who meet the eligibility criteria are randomly assigned to either an exercise intervention group or a control group. The intervention group performs a structured kettlebell-based exercise program three times per week for a duration of eight weeks, while the control group receives usual care without participation in the exercise program. Outcome measures are collected at baseline and after completion of the intervention period to evaluate changes associated with the exercise program.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males aged 18-25 years
2. Anterior pelvic tilt angle greater than 15°
3. Positive bilateral Thomas test
4. Observed mild hip flexion and knee flexion during standing posture
5. No history of spinal, pelvic, or lower limb surgeries

Exclusion Criteria:

1. Congenital anomalies of the lumbar vertebrae
2. Severe cardiovascular, neurological, or vascular diseases

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pelvic Tilt Angle | Baseline and 8 weeks after intervention
  Changes in pelvic tilt angle will be measured using the angle of the line connecting the Anterior Superior Iliac Spine (ASIS) and the Posterior Superior Iliac Spine (PSIS) relative to the horizontal, comparing pre- and post-intervention values between the exercise intervention group and the control group. The primary objective is to evaluate whether the kettlebell exercise program reduces the anterior pelvic tilt angle in male patients with Type A Lower Crossed Syndrome.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Physical Education, Hebei Normal University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.